CLINICAL TRIAL: NCT02791698
Title: The Accuracy of Late Night Urinary Free Cortisol/Creatinine and Hair Cortisol in Cushing's Syndrome Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, leonard.saiegh, Doctor, Bnai Zion Medical Center
Other Study IDs: 0049-15-BNZ
Record Dates: First submitted 2016-05-24; First posted 2016-06-07 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Cushing Syndrome
Keywords: cortisol; hair; urinary
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and hair
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will conduct a prospective study, in which they will determine sensitivity, specificity and diagnostic accuracy of late evening urinary free cortisol concentration/creatinine and hair cortisol in differentiating Cushing's syndrome from Pseudo-Cushing's syndrome.

DETAILED DESCRIPTION:
24h-Urine free cortisol (24h-UFC) and other screening tests may turn out normal in Cushing's syndrome (CS) patients, probably due to high variability and cyclicity in cortisol secretion. To rule out cyclic cortisol secretion, the recommendation is to repeat 24h-UFC measurements on different and several occasions. As 24h-UFC is technically inconvenient, especially in the elderly and in women, compliance may not be optimal, and results could be falsely low especially if collection is not properly conducted.

Alternatively, the status of cortisol circadian rhythm and urinary cortisol secretion may be assessed in a non-invasive and more convenient manner through the measurement of late evening urinary free cortisol concentration/creatinine concentration (Late-UFC). These measurements have been useful in screening outpatients for CS, but their performances have not been properly and enough validated.

It appears that the assessment of Late-UFC can offer a non-invasive and convenient diagnostic tool for evaluating cortisol circadian rhythm and urinary cortisol secretion in ambulatory populations, especially in the case of patients for whom 24h-UFC should be repeated yet is technically not convenient to perform.

Hair sample testing has gained increasing attention and recognition over the last 20 years, especially for detecting illegal drug use and for other forensic purposes. This is because hair provides a relatively long-term retrospective record of levels of various bio-markers in the body.

In light of the foregoing evidence, it has been suggested that hair cortisol measurement could be a novel method for assessing dynamic systemic cortisol exposure, and could provide unique historical information on variation and cyclicity in cortisol exposure.

The investigators will conduct a prospective cohort study which will include patients referred to outpatient endocrinology clinic for medical evaluation due to CS suspicion or adrenal incidentaloma evaluation. Participants will be asked to provide informed consent before study enrollment. All Participants will be asked to perform the routine screening tests for CS diagnosis. On the same day participants will collect the 24h-UFC, they will be asked to empty their urinary bladder at 22:00 hour to the urinary collection bottle, and to give a single urinary sample at 24:00 hour for Late-UFC determination.

Immediately after study enrollment, hair sample of approximately 100-150 strands and 2-3 cm long will be collected from the posterior vertex, and cortisol concentration in hair will be determined.

All patients enrolled will be diagnosed as "CS", "Pseudo-Cushing's syndrome" or "undermined". CS will be classified as ACTH-dependent CS or ACTH-independent CS. ACTH-dependent CS will be diagnosed when at least two screening tests for CS are positive (not including Late-UFC and HC), normal or elevated basal plasma ACTH concentration, and positive ACTH stained histology and/or post-surgical hypoadrenalism. ACTH-independent CS will be diagnosed when at least one screening test is positive, depressed basal plasma ACTH concentration (ACTH concentration below 2.2 pmol/L) and the patient has adrenal-post-surgical hypoadrenalism. Patients will be diagnosed as "Pseudo-Cushing's syndrome" when only one screening test is positive out of at least three tests performed, patients harboring no typical features for CS, and there is no deterioration in biochemical or clinical status during the study follow-up. Patients will be diagnosed as "undermined" when harboring two or more positive screening tests, yet the clinical and biochemical profile do not support definitive diagnosis.

To address the questions of the study, the investigators will compare the two groups of "CS" and "Pseudo-Cushing's syndrome" determining sensitivity, specificity and diagnostic accuracy of Late-UFC and Hair cortisol in differentiating Cushing's syndrome from Pseudo-Cushing's syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to our outpatient endocrinology clinic for medical evaluation due to CS suspicion or adrenal incidentaloma evaluation

Exclusion Criteria:

1. Serum creatinine level concentration above 1.5 mg/deciliter
2. Systemic, dermal or nasal steroid use
3. Chronic inflammatory disease
4. Any infectious disease requiring hospitalization or more that 2 weeks of antibiotic treatment in the previous 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred to our outpatient endocrinology clinic for medical evaluation due to Cushing's syndrome suspicion or adrenal incidentaloma evaluation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Cushing's syndrome | 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saiegh, M.D., Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Saiegh leonard, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No